CLINICAL TRIAL: NCT02465554
Title: Imaging and Omics for Cardiovascular Risk During NASA Deep Space Missions
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Jonathan R. Lindner, MD, Professor, Oregon Health and Science University
Other Study IDs: IRB00011874
Record Dates: First submitted 2015-06-03; First posted 2015-06-08 (Estimated); Last update posted 2018-01-12 (Actual); Status verified 2018-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- No atherosclerosis cohort: This group will have patients who have undergone clinically-indicated CT coronary angiography (CT-A) and who have no plaque and an Agatston score of "0". They will then undergo a myocardial contrast echocardiography study during vasodilator stress to subdivide risk further into "No atherosclerosis/endothelial function normal" and "No atherosclerosis/endothelial function abnormal". Blood will then be collected for metabolomics, lipidomic and whole genome sequencing.
  Interventions: Procedure: Myocardial contrast echocardiography
- Atherosclerosis cohort: This group will have patients who have undergone clinically-indicated CT coronary angiography (CT-A) and who have non-critical plaque (<50% diameter) and at least 1 high risk feature according to the ROMICAT indices. They will then undergo a myocardial contrast echocardiography study during vasodilator stress to subdivide risk further into "atherosclerosis/endothelial function normal" and "atherosclerosis/endothelial function abnormal". Blood will then be collected for metabolomics, lipidomic and whole genome sequencing.
  Interventions: Procedure: Myocardial contrast echocardiography

INTERVENTIONS:
Procedure: Myocardial contrast echocardiography — Myocardial contrast echocardiography will be performed to further stratify risk as described in the cohort section.

SUMMARY:
The purpose of this study is to develop new approaches for screening astronauts for cardiovascular risk during deep space missions.

DETAILED DESCRIPTION:
The purpose of this study is to develop new approaches for screening astronauts for cardiovascular risk during deep space missions. In this protocol, two different forms of imaging will be used to evaluate coronary plaque development (CT coronary angiography) and microvascular function (myocardial contrast echocardiography) to stratify CV risk. Based on this stratification, "omic" patterns (targeted metabolomics, lipidomic, and whole genome sequencing) will be assessed to determine whether there are any patterns that can add to existing predictive models. Outcomes measures will involve correlation of "omic" patterns to incremental risk scaling from lowest (no plaque and normal endothelial function) to highest (+ plaque and endothelial dysfunction).

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for clinically indicated CT coronary angiography within 6 months
* No obstructive coronary plaque and an Agatston score of 0 or At least one obstructive coronary plaque <50% diameter and one other high risk feature on CT-A (positive remodeling, scattered calcification, low Hounsfield units, or "napkin ring" sign.

Exclusion Criteria:

* Known CAD or other atherosclerotic disease
* Valvular heart disease (moderate or more) and congenital heart disease
* Heart failure
* Pregnancy
* Allergy to ultrasound contrast agent.
* Right to left shunt

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients referred for clinically-indicated CT coronary angiography.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-09; Primary Completion 2017-12-31 (Actual); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Omic patterns of atherosclerosis | 2 weeks
  In this study, "outcomes" are essentially pre-determined by the patient population according to imaging stratification. Omic patterns of will be assessed by advanced informatics modeling (Random Forest analysis) to determine metabolomic, genomic, and lipidomic patterns that vary according to incremental risk scaling from lowest (no plaque and normal endothelial function) to highest (+ plaque and endothelial dysfunction).

CONTACTS AND LOCATIONS:
Locations (1):
- Oregon Health & Science University, Portland, Oregon, United States